CLINICAL TRIAL: NCT00005822
Title: A Phase I Pharmacokinetic, Pharmacodynamic, and Clinical Study of the Combination of the Angiogenesis Inhibitor SU5416 and Doxorubicin in Inflammatory Breast Cancer
Brief Title: SU5416 and Doxorubicin in Treating Patients With Stage IIIB or Stage IV Inflammatory Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Beth A. Overmoyer, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU5199; U01CA062502 (NIH); P30CA043703 (NIH); CWRU-5199; NCI-T99-0099
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; stage IIIB breast cancer; inflammatory breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms; Breast Neoplasms, Male | interventions — Doxorubicin; Semaxinib; Radiotherapy; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: doxorubicin hydrochloride — Patients receive doxorubicin IV continuously over 72 hours on days 1-3 of course 1. For all subsequent courses, patients receive doxorubicin as in course 1. Treatment repeats every 21 days for 5 courses in the absence of disease progression or unacceptable toxicity.
Drug: semaxanib — For all subsequent courses, after course 1 patients SU5416 IV over 1 hour twice weekly (on days 1 and 4) beginning on week 2 of course 2. Treatment repeats every 21 days for 5 courses in the absence of disease progression or unacceptable toxicity.
  Other Names: SU5416
Procedure: conventional surgery — Patients undergo a modified radical mastectomy.
Radiation: radiation therapy — Patients undergo radiotherapy to the chest wall and regional lymph nodes.
Drug: tamoxifen — Patients with estrogen or progesterone receptor positive disease receive oral tamoxifen for 5 years after radiotherapy.

SUMMARY:
RATIONALE: SU5416 may stop the growth of breast cancer by stopping blood flow to the tumor. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining SU5416 with chemotherapy may kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of combining SU5416 and doxorubicin in treating patients who have stage IIIB or stage IV inflammatory breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of SU5416 and doxorubicin in patients with stage IIIB or IV inflammatory breast cancer.
* Determine the overall response, response rate, and progression-free survival rate of patients treated with this regimen.
* Determine the antiangiogenic effects of this regimen in these patients.
* Assess the relationship of plasma levels of these drugs with safety and efficacy in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive doxorubicin IV continuously over 72 hours on days 1-3 of course 1. For all subsequent courses, patients receive doxorubicin as in course 1 and SU5416 IV over 1 hour twice weekly (on days 1 and 4) beginning on week 2 of course 2. Treatment repeats every 21 days for 5 courses in the absence of disease progression or unacceptable toxicity. After chemotherapy, all patients undergo a modified radical mastectomy and radiotherapy to the chest wall and regional lymph nodes. Patients with estrogen or progesterone receptor positive disease receive oral tamoxifen for 5 years after radiotherapy.

Cohorts of 3-6 patients receive escalating doses of SU5416 and doxorubicin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, an additional 3 patients may be treated at that dose level.

Patients are followed every 3 months until disease progression.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study within 6-9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage IIIB or IV (supraclavicular lymph node involvement or metastasis) inflammatory breast cancer

  * Primary or secondary
* No brain metastases or primary brain tumors
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Male or female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* WBC at least 3,500/mm^3
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin greater than 9.0 g/dL

Hepatic:

* Bilirubin normal
* AST and ALT less than 2 times upper limit of normal
* PT and PTT normal OR
* INR less than 1.1

Renal:

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* LVEF at least 50% by MUGA
* No New York Heart Association class III or IV heart disease
* No uncompensated coronary artery disease
* No myocardial infarction or unstable angina within the past 6 months
* No deep venous or arterial thrombosis within the past 3 months

Pulmonary:

* No history of pulmonary embolism within the past 3 months

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of diabetes mellitus with severe peripheral vascular disease
* No other prior or concurrent malignancies within the past 10 years except inactive nonmelanomatous skin cancer or carcinoma in situ of the cervix
* No other uncontrolled illnesses

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent epoetin alfa or filgrastim (G-CSF)

Chemotherapy:

* No more than 2 prior chemotherapy regimens allowed
* No prior doxorubicin or other anthracycline

Endocrine therapy:

* Not specified

Radiotherapy:

* Prior radiotherapy allowed

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2000-04; Primary Completion 2002-12 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of SU5416 and doxorubicin in patients with stage IIIB or IV inflammatory breast cancer. | Treatment repeats every 21 days for 5 courses in the absence of disease progression or unacceptable toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Beth A. Overmoyer, MD, FACP, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Cleveland, Ohio, United States